CLINICAL TRIAL: NCT04131868
Title: The Contribution of Stressful Life Events and Insufficient Sleep to Reward-Related Brain Function and Depression in Adolescent Girls
Brief Title: Sleep and Girls' Emotions Study
Acronym: SAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Melynda Casement, Assistant Professor, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: K01MH103511 (NIH)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended sleep opportunity (Experimental)
  Interventions: Behavioral: Extended sleep opportunity
- Typical sleep opportunity (Active Comparator)
  Interventions: Behavioral: Typical sleep opportunity

INTERVENTIONS:
Behavioral: Typical sleep opportunity — Typical sleep opportunity with consistent sleep timing for 1 week
  Arms: Typical sleep opportunity
Behavioral: Extended sleep opportunity — Extended sleep opportunity by 90 min per night with consistent sleep timing for 1 week
  Arms: Extended sleep opportunity

SUMMARY:
This study evaluates whether increasing sleep duration can increase neural and behavioral response to rewards and decrease depressive symptoms in 18- to 22-year-old women with insufficient sleep and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Insufficient sleep (total sleep time < 8 hours per night, with sleepiness scores ≥ 6 on the Epworth Sleepiness Scale OR ≥ 16 on the PROMIS Sleep Related Impairment Scale)
* Symptoms of depression (≥ 15 on the Center for Epidemiological Studies for Depression Scale)

Exclusion Criteria:

* Current insomnia, hypersomnia, sleep disordered breathing, sleep movement disorder, or circadian rhythm disorder
* History of head injury with loss of consciousness within the past two years
* History of head injury with loss of consciousness two or more years ago and meet criteria for post concussion syndrome
* Neurological disorder
* Use of psychiatric medications
* Current psychotic symptoms
* Active suicidal ideation
* Conditions that are contraindicated for MRI (e.g., ferromagnetic material in the body)
* Meet criteria for current substance use disorder with greater than mild severity

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 34 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 1 week
  Center for Epidemiological Studies Depression Scale score. The CESD-R is a 20-item measure of the frequency of depressive symptoms, with each item rated on a scale from 0 (not at all or less than one day) to 5 (nearly every day). Total scores range from 0 to 100, with higher scores indicating greater number and frequency of depressive symptoms.
Reward-related brain function | 1 week
  BOLD fMRI response during Reward Guessing Task
Sleep duration | 1 week
  Mean actigraphy-measured sleep duration

SECONDARY OUTCOMES:
Positive affect | 1 week
  International Positive and Negative Affect Scale Short Form - Positive Affect score. The I-PANAS-SF is a 10-item scale that asks participants to rate the extent to which 5 positive and 5 negative adjectives describe them on a scale of 1 (never) to 5 (always). Scores for each positive adjective are summed to produce a Positive Affect (PA) score ranging from 5 to 25, with higher scores indicating more positive affect.
Negative affect | 1 week
  International Positive and Negative Affect Scale Short Form - Negative Affect score. The I-PANAS-SF is a 10-item scale that asks participants to rate the extent to which 5 positive and 5 negative adjectives describe them on a scale of 1 (never) to 5 (always). Scores for each negative adjective are summed to produce a Negative Affect (PA) score ranging from 5 to 25, with higher scores indicating more negative affect.
Reward effort | 1 week
  Effort Expenditure for Rewards Task score
Reward-related functional connectivity | 1 week
  BOLD fMRI psychophysiological striatal-medial prefrontal cortex interaction

CONTACTS AND LOCATIONS:
Overall Officials: Melynda D Casement, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided